CLINICAL TRIAL: NCT00559039
Title: Fetal, Infant and Early Childhood Antecedents of Cancer in Women: Maternal Cohort Study of the Nurses' Health Studies
Brief Title: Effects of Fetal, Infant, and Early Childhood Exposures on Adult Cancer Risk in Women
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: 999901015; 01-C-N015; CDR0000565931; NCT00340145 (obsolete NCT alias)
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: breast cancer; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Other: questionnaire administration
Procedure: evaluation of cancer risk factors

SUMMARY:
RATIONALE: Gathering information about pregnancy, infancy, and early childhood exposures may help doctors identify cancer risk factors, and may help the study of cancer.

PURPOSE: This natural history study is looking at the effects of fetal, infant, and early childhood exposures on adult cancer risk in women.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if fetal, infant, and early childhood exposures are associated with adult cancer risk in women.

OUTLINE: Mothers of nurses complete questionnaires to collect maternal data, such as pregnancy weight gain, diet during pregnancy, maternal pre-eclampsia, gestational diabetes, gestational age at birth, birth weight, and infant feeding practices. Maternal data is linked to other data collected from critical time periods in the nurses's life cycle, such as menarche, first pregnancy, or adult dietary intake.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Mother of a nurse who is a participant in the Nurses' Health Studies I and II

  * Nurse free of cancer in the year 2000

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128700 (Estimated)
Dates: Start 2000-10; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Diagnosis of incident cancers and other chronic diseases
Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Michele R. Forman, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States